CLINICAL TRIAL: NCT00505089
Title: An Exploratory, Open Label Pharmacokinetic - Pharmacodynamic Study to Compare Subcutaneous Versus Intravenous Administration of ACZ885 in Adult Patients With Established Rheumatoid Arthritis
Brief Title: Efficacy and Safety of Subcutaneous Versus Intravenous ACZ885 in Adult Patients With Established Rheumatoid Arthritis
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CACZ885A2206
Record Dates: First submitted 2007-07-19; First posted 2007-07-20 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Rheumatoid Arthritis
Keywords: pharmacokinetic, pharmacodynamic, subcutaneous, intravenous, ACZ885, patients, rheumatoid, arthritis.
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis | interventions — canakinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): ACZ885 10mg/kg subcutaneous
  Interventions: Drug: ACZ885
- 2 (Experimental): ACZ885 5mg/kg intravenous
  Interventions: Drug: ACZ885
- 3 (Experimental): ACZ885 2mg/kg subcutaneous
  Interventions: Drug: ACZ885
- 4 (Experimental): ACZ885 1mg/kg intravenous
  Interventions: Drug: ACZ885

INTERVENTIONS:
Drug: ACZ885
  Arms: 1
Drug: ACZ885
  Arms: 2
Drug: ACZ885
  Arms: 3
Drug: ACZ885
  Arms: 4

SUMMARY:
This study will investigate the pharmacokinetic (PK) / total IL-1beta pharmacodynamic (PD) relationship in joint fluids of patients with rheumatoid arthritis (RA) treated with different doses of ACZ885 and to evaluate the impact of the subcutaneous (s.c.) versus intravenous (i.v.) route of administration.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 - 75 years (inclusive).
* Body weight must be between 50 and 100 kg (inclusive).
* Post-menopausal or surgically sterile female patients. Women of child-bearing potential if already on a stable dose of methotrexate and are practicing effective contraception for at least 3 months prior to screening, have a negative pregnancy test at screening and baseline, and are willing to use 2 forms of contraception including at least 1 barrier method during the study and for at least 2 months following the completion/discontinuation of the study. Male patients must be willing to use an effective contraception method during the study and at least for 2 months following the completion/discontinuation of the study.
* Diagnosis of Rheumatoid Arthritis, classified by ARA (American Rheumatism Association) 1987 revised criteria (Appendix 2). Disease duration of at least 6 months prior to randomization is essential.
* Functional status class I, II or III classified according to the ACR (American College of Rheumatology) 1991 revised criteria (Appendix 3).
* Active disease at screening and baseline (Day 1 predose) evaluation (same evaluator): ≥ 6 tender and ≥ 6 swollen joints of 28 examined (including any effused joint) and either a) Westergren erythrocyte sedimentation rate (ESR) ≥ 28 mm/hour, or b) C-reactive protein (CRP) ≥ 1.0 mg/dL.
* Prior treatment with 1-3 disease-modifying anti-rheumatic drugs (DMARDs) - Patients should have failed at least 1 DMARD but should not be deemed "refractory to all therapies". Patients should be on a current treatment with methotrexate ≤ 25 mg/week and with the current dose stable for at least 3 months. All patients will take folic acid 1 mg daily, or 5 mg weekly post MTX dose, to minimize toxicity, according to local guidelines. In addition to methotrexate, patients may be on either a stable dose of non-steroidal anti-inflammatory drugs (NSAIDs) and/or a stable dose of oral corticosteroids (prednisone or equivalent ≤ 10 mg daily) for at least 4 weeks prior to randomization. Patients who failed any DMARDs will be allowed.
* Negative purified protein derivative (PPD) tuberculin skin test reaction (PPD 5 tuberculin units or as according to local standard practice).
* Patients with a total white cell count and platelet count clinically acceptable for patients with RA; hemoglobin must be ≥ 10 g/dL and hematocrit ≥ 30% at screening and baseline.

Exclusion Criteria:

* Previous treatment with anti-TNF-α or anti IL-1 therapy (or other biological therapy), immunosuppressive agents such as cyclosporine, mycophenolate or tacrolimus. The following washout period will be required for such patients to be eligible to participate in the trial.

  1. 2 months washout prior to screening for etanercept or adalimumab
  2. 3 months washout prior to screening for infliximab
  3. 3 months washout prior to screening for rituximab
  4. 1 month washout prior to screening for cyclosporine, mycophenolate and tacrolimus.
* If patient has been discontinued from other DMARDs for lack of efficacy or toxicity, the patient should be at least 1 month off the agent and the effects of that agent should have dissipated according to the recognized duration of effect (e.g., sulfasalazine, hydroxychloroquine), or standard washout procedure (cholestyramine for leflunomide). Importantly, discontinuation should not be undertaken only for the purposes of participation in this study.
* Patients who have received intra-articular or systemic corticosteroid injections having been required for treatment of acute RA flare (not being part of a regular therapeutic regimen) within four weeks prior to randomization.
* Presence of or history of Major chronic inflammatory autoimmune diseases like psoriasis, psoriatic arthritis, spondyloarthropathy, inflammatory bowel disease or systemic lupus erythematosus.

Renal trauma, glomerulonephritis or patient with one kidney. Patients with congestive heart failure (New York Heart Association class > III), QT prolongation syndrome or poorly controlled diabetes mellitus. Patients with a history of QTc prolongation will be excluded. A positive HIV test result, Hepatitis B surface antigen or Hepatitis C test result. Significant illness within 2 weeks prior to dosing or any active systemic infection or medical condition that may require treatment or therapeutic intervention during the study. Hypersensitivity to any biological agents, serious allergic reaction, collagen disease, neurological disease (including demyelinating disease). Any joint surgery in past 8 weeks or planned surgery within next 5 months. Cancer (other than basal cell cancer or adequately treated carcinoma-in-situ of the cervix). Drug or alcohol abuse within the 12 months prior to dosing or evidence of such indicated by the laboratory assays conducted during the screening or baseline evaluations. Underlying metabolic, endocrine, hematologic, pulmonary, cardiac, blood, renal, hepatic, infectious, psychiatric or gastrointestinal conditions which places the patient at unacceptable risk for participation in a study of an immunomodulatory therapy.

* Treatment with an investigational agent within 12 weeks prior to enrollment or longer if required by local regulation.
* Pregnant or breastfeeding women.
* Donation or loss of 400 mL or more of blood within 8 weeks prior to dosing

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-08; Primary Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
- Pharmacokinetic/total IL-1beta pharmacodynamic relationship in joint fluids of patients with rheumatoid arthritis treated with different doses of ACZ885 - Impact of the subcutaneous versus intravenous administration | End of study

SECONDARY OUTCOMES:
- PK/PD of ACZ885 in patient serum and to evaluate impact of s.c. versus i.v. administration - Efficacy via response to treatment (ACR 20% improvement [ACR 20],50,70 & 90) | Days 8,15,29,43 and study completion

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigative site
Locations (9):
- Belgium (2):
  - Novartis Investigative site, Antwerp
  - Novartis Investigator Site, Liège
- Germany (4):
  - Novartis Investigative site, Berlin
  - Novartis Investigator Site, Berlin
  - Novartis Investigator Site, Hanover
  - Novartis Investigator Site, Leipzig
- Novartis investigative site, Leiden, Netherlands
- Poland (2):
  - Novartis Investigative Site, Grodzisk Mazowiecki
  - Novartis Investigator Site, Poznan